CLINICAL TRIAL: NCT04435574
Title: Comparison of Lactoferrin vs Traditional Iron Therapy for Treatment of Iron Deficiency Anemia in School-age Children.
Brief Title: Lactoferrin for Treatment of Iron Deficiency Anemia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Saeed Salah Abduljalil Soliman, Lecturer of family medicine, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70777
Record Dates: First submitted 2018-08-31; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: the population for the study will be Scholar age Children attend family medicine clinic for treatment of iron deficiency anemia and their parents accept participation in the study.
  For confirmation of the diagnosis of iron deficiency anemia the following investigations will be done:
  * CBC
  * Serum total iron
  full medical history and examination will be performed. study participants will be assigned to either group A (lactoferrin group) or group B (ferrous sulfate group), and will receive the corresponding medication for 8 weeks.
  4 weeks follow up for side effects and hemoglobin level and 8 weeks follow up for side effects, hemoglobin level and serum iron will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): group A is lactoferrin group, receiving 100mg sachet of lactoferrin once daily.
  Interventions: Drug: Lactoferrin
- Group b (Active Comparator): group B is the ferrous sulfate group, receiving 6mg/kg/ day single dose of ferrous sulfate.
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Lactoferrin — Bovine Lactoferrin 100mg sachets.
  Arms: Group A
Drug: Ferrous Sulfate — 6mg/kg of ferrous sulfate.
  Arms: Group b

SUMMARY:
Anemia is a great public health problem affecting both developing and developed countries. Iron deficiency anemia represents about 50% of causes of anemia worldwide.

Lactoferrin fortified milk has a positive effect on Hb and iron status of infants.

the hypothesis of this study is "lactoferrin may have comparable efficacy to ferrous sulfate therapy with more tolerability and fewer side effects".

the research question of this study is whether oral lactoferrin is effective for treatment of iron deficiency anemia, compared to traditional ferrous sulfate therapy regarding hemoglobin rise and side effects and tolerability.

DETAILED DESCRIPTION:
Anemia is a great public health problem affecting both developing and developed countries. It is considered the most prevalent form of malnutrition in children and adolescents.

Supplementation with standard iron therapy is the main treatment of iron deficiency anemia.

There are two types of iron that are available: ferric and ferrous iron but ferrous iron better in absorption so it is more common in use.

Three types of ferrous iron are present: ferrous sulfate, ferrous fumarate, and ferrous gluconate but all forms have annoying gastrointestinal side effects including diarrhea, anorexia, heartburn, vomiting, nausea, abdominal cramps, upset stomach, and constipation making continuation on it for many weeks unpleasant for all even adults.

Studies have been performed to explore the effect of oral bovine lactoferrin on iron absorption on pregnant women. Many studies showed that oral bovine lactoferrin for pregnant women increased levels of hemoglobin, total serum iron, and ferritin and decreased the prevalence of iron deficiency anemia. although ferrous sulfate and lactoferrin both of them significantly improve the body's iron stores to the same extent, gastrointestinal side effects of lactoferrin were extremely lower than that of ferrous sulfate so oral bovine lactoferrin can replace iron forms in the treatment of iron deficiency anemia in pregnancy.

Lactoferrin is a glycoprotein from the transferrin family consist of 691 amino acids. It is a component of exocrine secretions such as milk and saliva and is present in neutrophil granules. Lactoferrin was identified in 1939 in bovine milk and isolated in 1960 from both human and bovine milk. Human colostrum shows the highest levels of lactoferrin while mature milk and other secretions present lower.

Lactoferrin was used in children as antimicrobial in cases of acute diarrhea.In vitro data document the growth inhibition of the diarrheal associated organisms: rotavirus, cholera, salmonella, and shigella by human lactoferrin.

Studies about Milk formula fortified with bovine lactoferrin confirmed its positive effect on Hb and iron status of infants. Recombinant human lactoferrin was extracted from rice seed, is used by Ventria Bioscience as a dietary supplement for treatment of iron of deficiency anemia.

Rationale:

Iron deficiency anemia has a high prevalence rate in scholar age children with their big need to iron for anabolic processes of growth. Supplementation with standard iron therapy is the main treatment however its unpleasant side effects negatively affect patient compliance.

Hypothesis:

Lactoferrin may have a positive effect in the treatment of iron deficiency anemia in school-age children. Lactoferrin side effects less than standard iron therapy.

Research question:

Is lactoferrin usage in the treatment of iron deficiency anemia in scholar age children has a positive effect and little side effects in comparison with standard iron therapy (ferrous sulfate)?.

1. Objectives

This study aims to:

1. Evaluation of the effect of oral lactoferrin in the treatment of iron deficiency anemia in school-age children in comparison with standard iron therapy (ferrous sulfate).
2. Assessment of side effects occurs with the usage of lactoferrin.

ELIGIBILITY:
Inclusion Criteria:

* Children with iron deficiency anemia.

Exclusion Criteria:

* Malabsorption diseases as coeliac disease.
* Diseases causing chronic blood loss as Meckel diverticulum.
* Documented history of allergy to lactoferrin or ferrous sulfate.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 8 weeks
  hemoglobin%
Total serum iron | 8 weeks
  Total serum iron

SECONDARY OUTCOMES:
Side effects profile | 4 weeks
  Score of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Khfaji, Associate professor, Principal Investigator — Cairo University
Locations (1):
- Primary care center, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stoltzfus R. Defining iron-deficiency anemia in public health terms: a time for reflection. J Nutr. 2001 Feb;131(2S-2):565S-567S. doi: 10.1093/jn/131.2.565S. PMID 11160589
- [Background] Paesano R, Torcia F, Berlutti F, Pacifici E, Ebano V, Moscarini M, Valenti P. Oral administration of lactoferrin increases hemoglobin and total serum iron in pregnant women. Biochem Cell Biol. 2006 Jun;84(3):377-80. doi: 10.1139/o06-040. PMID 16936810
- [Background] Paesano R, Pietropaoli M, Gessani S, Valenti P. The influence of lactoferrin, orally administered, on systemic iron homeostasis in pregnant women suffering of iron deficiency and iron deficiency anaemia. Biochimie. 2009 Jan;91(1):44-51. doi: 10.1016/j.biochi.2008.06.004. Epub 2008 Jun 14. PMID 18601971
- [Background] Rezk M, Dawood R, Abo-Elnasr M, Al Halaby A, Marawan H. Lactoferrin versus ferrous sulphate for the treatment of iron deficiency anemia during pregnancy: a randomized clinical trial. J Matern Fetal Neonatal Med. 2016;29(9):1387-90. doi: 10.3109/14767058.2015.1049149. Epub 2015 Jun 3. PMID 26037728